CLINICAL TRIAL: NCT05906940
Title: Effects of Transcutaneous Auricular Vagus Nerve Stimulation on Basic Autonomic Nervous System Activity
Brief Title: Vagus Nerve Stimulation for Autonomic Nervous System Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Alper Percin, Principal Investigator, Bahçeşehir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AP0005
Record Dates: First submitted 2023-05-29; First posted 2023-06-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Autonomic Nervous System Imbalance
Keywords: Autonomic Nervous Systems; Vagal Nerve Stimulation; Heart Rates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Participants (Experimental): Participants in this group will be measured heart rate variability before and after transcutaneous vagus nerve stimulation.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation — As a vagus stimulation protocol, bilateral auricular stimulation and stimulation frequency of 10 Hz, pulse width of 300 µs, biphasic application for 20 minutes, each participant will be stimulated twice, with at least 48 hours between them.

SUMMARY:
There are no generally accepted values for transcutaneous vagus nerve stimulation (taVSS application parameters (amplitude, frequency, intensity, duration, side) yet, therefore there are heterogeneous applications in studies. Although positive effects have been shown in different neurological, psychiatric and musculoskeletal diseases, taVSS treatment is not available yet. It is not clear which parameters are important in patient selection.In this study, it was aimed to investigate the change of taVSS effect in healthy individuals according to the level of autonomic nervous system activity before stimulation.

DETAILED DESCRIPTION:
Healthy individuals between the ages of 18-45 without any disease will be included in the study. Male and female participants will be included in the study. Heart rate variability will be measured after participants are included in the study. A short 5-minute measurement will be made with the Polar H7 device, which can be measured with the belt attached to the chest. Heart Rate Variability measurement will be analyzed with the Kubios HRV program. Participants will be distributed to groups according to the SNS index and PNS index values obtained as a result of the Kubios analysis. According to the index scores obtained, the distribution of the groups will be made as <-2, between -2 and +2 and >2. Afterwards, 20 minutes of taVSS stimulation will be performed. As a vagus stimulation protocol, bilateral auricular stimulation and stimulation frequency of 10 Hz (Heartz), pulse width of 300 µs (microseconds) for 20 minutes, biphasic application will be given to each participant 2 times, with at least 48 hours between them.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between the ages of 18-45 will be included in the study.

Exclusion Criteria:

* Having an acute or chronic disease,
* Having previously undergone transcutaneous vagus nerve stimulation,
* Not smoking or using alcohol,
* Being in the post-menopausal stage in women,
* Being in the post-andropausal period in men,
* Being on constant medication,
* In menstruating women, stimulation and heart rate assessment will be postponed to the next week.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability Parameters-Stress Index | 5 minutes (short measurement) measurement of heart rate variability
  Stress index which is a geometric measure of HRV reflecting cardiovascular system stress. High values of SI indicate reduced variability and high sympathetic cardiac activation.
Heart Rate Variability Parameters-RMSSD | 5 minutes (short measurement) measurement of heart rate variability
  RMSSD is a measure of short-term (beat-by-beat) variability. It equals the root mean square of successive differences.
Heart Rate Variability Parameters-LF (Low Frequency) | 5 minutes (short measurement) measurement of heart rate variability
  Power in the Low Frequency band of the HRV spectrum, often between 0.04 - 0.15 Hz, often reported in units of milliseconds-squared.
Heart Rate Variability Parameters-HF (High Frequency) | 5 minutes (short measurement) measurement of heart rate variability
  Power in the High Frequency band of the HRV spectrum, often between 0.15-0.40 Hz, often reported in units of milliseconds-squared.
Heart Rate Variability Parameters-LF/HF Ratio | 5 minutes (short measurement) measurement of heart rate variability
  LF/HF Ratio: A ratio of Low Frequency to High Frequency.
Heart Rate Variability Parameters-SNS Index | 5 minutes (short measurement) measurement of heart rate variability
  Sympathetic cardiac activity is known to 1) increase heart rate, 2) decrease HRV, reducing especially quick RSA related changes in RR interval, and 3) increase the ratio between lower frequency and higher frequency oscillations in HRV data
Heart Rate Variability Parameters-PNS Index | 5 minutes (short measurement) measurement of heart rate variability
  Parasympathetic cardiac activity is known to 1) decrease heart rate (i.e. increase the time interval between successive heart beats), 2) increase HRV via enhanced respiratory sinus arrhythmia (RSA) component (i.e. increasing the quick changes in RR interval linked to respiration - shortening of RR intervals during inhalation and lengthening of RR intervals during exhalation), and 3) decrease the ratio between lower frequency and higher frequency oscillations in HRV time series (i.e. increase the relative amount of quick RSA originated fluctuations in HRV compared to slower short-term fluctuations)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Veysel Özden, MD, PhD., Study Director — Iğdır University Physiotherapy and Rehabilitation Laboratory
Locations (1):
- Iğdır University, Iğdır, Iğdır Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ben-Menachem E, Revesz D, Simon BJ, Silberstein S. Surgically implanted and non-invasive vagus nerve stimulation: a review of efficacy, safety and tolerability. Eur J Neurol. 2015 Sep;22(9):1260-8. doi: 10.1111/ene.12629. Epub 2015 Jan 23. PMID 25614179
- [Result] Milby AH, Halpern CH, Baltuch GH. Vagus nerve stimulation for epilepsy and depression. Neurotherapeutics. 2008 Jan;5(1):75-85. doi: 10.1016/j.nurt.2007.10.071. PMID 18164486
- [Result] Butt MF, Albusoda A, Farmer AD, Aziz Q. The anatomical basis for transcutaneous auricular vagus nerve stimulation. J Anat. 2020 Apr;236(4):588-611. doi: 10.1111/joa.13122. Epub 2019 Nov 19. PMID 31742681